CLINICAL TRIAL: NCT02429557
Title: Hemodynamic Mechanisms of Abdominal Compression in the Treatment of Orthostatic Hypotension in Autonomic Failure
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Luis E Okamoto, Research Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 140634; 1R01HL144568-01A1 (NIH)
Record Dates: First submitted 2015-04-21; First posted 2015-04-29 (Estimated); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Orthostatic Hypotension; Pure Autonomic Failure; Multiple System Atrophy; Autonomic Failure
Keywords: autonomic failure; orthostatic hypotension; compression garments; treatment
MeSH Terms: conditions — Hypotension, Orthostatic; Pure Autonomic Failure; Multiple System Atrophy | interventions — Midodrine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Abdominal compression and placebo pill (Experimental): Abdominal compression with an inflatable abdominal binder (up to 40 mmHg) during head up tilt, and placebo pill given 1 hour before the second head up tilt
  Interventions: Other: Abdominal compression; Drug: Placebo pill
- Sham abdominal compression and placebo (Sham Comparator): Sham abdominal compression with an inflatable abdominal binder (~5 mmHg) during head up tilt, and placebo pill given 1 hour before the second head up tilt
  Interventions: Other: Sham abdominal compression; Drug: Placebo pill
- Abdominal compression and midodrine (Experimental): Abdominal compression with an inflatable abdominal binder (up to 40 mmHg) during head up tilt, and midodrine 2.5-10 mg PO given 1 hour before the second head up tilt
  Interventions: Other: Abdominal compression; Drug: midodrine
- Sham abdominal compression and midodrine (Active Comparator): Sham abdominal compression with an inflatable abdominal binder (~5 mmHg) during head up tilt, and midodrine 2.5-10mg PO given 1 hour before the second head up tilt
  Interventions: Other: Sham abdominal compression; Drug: midodrine

INTERVENTIONS:
Other: Abdominal compression — Abdominal compression of 40 mmHg with a commercial inflatable cuff applied during head up tilt
  Other Names: abdominal binder
  Arms: Abdominal compression and midodrine; Abdominal compression and placebo pill
Other: Sham abdominal compression — Sham abdominal compression of 5 mmHg with a commercial inflatable cuff applied during head up tilt
  Other Names: abdominal binder
  Arms: Sham abdominal compression and midodrine; Sham abdominal compression and placebo
Drug: Placebo pill — Placebo pill given 1 hour before the second heat up tilt
  Arms: Abdominal compression and placebo pill; Sham abdominal compression and placebo
Drug: midodrine — Midodrine single dose 2.5-10mg PO given 1 hour before the second head up tilt
  Other Names: ProAmatine
  Arms: Abdominal compression and midodrine; Sham abdominal compression and midodrine

SUMMARY:
Compression garments have been shown to be effective in the treatment of orthostatic hypotension in autonomic failure patients. The purpose of this study is to determine the hemodynamic mechanisms by which abdominal compression (up to 40 mm Hg) improve the standing blood pressure and orthostatic tolerance in these patients, and to compare them with those of the standard of care midodrine. The investigators will test the hypothesis that abdominal compression will blunt the exaggerated fall in stroke volume and the increase in abdominal vascular volume during head up tilt.

DETAILED DESCRIPTION:
Patients with autonomic failure are characterized by disabling orthostatic hypotension (low blood pressure on standing) due to severe impairment of the autonomic nervous system. Compression garments such as waist-high stockings and abdominal binders have been shown to improve orthostatic hypotension in these patients. The purpose of this study is to determine the hemodynamic mechanisms by which abdominal compression (up to 40 mm Hg) improve the standing blood pressure and orthostatic tolerance in these patients, and to compare them with those of the standard of care midodrine. The investigators will test the hypothesis that abdominal compression will blunt the exaggerated fall in stroke volume and the increase in abdominal vascular volume during head up tilt. This study will help us better understand the contribution of the abdominal veins to orthostatic hypotension and the mechanisms underlying this non-pharmacological therapeutic approach.

Participants will be studied in a tilt table in two separate days in a randomized, crossover fashion with sham abdominal compression (~5 mmHg) and active compression (~40 mmHg).

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients,
* between 18-80 yrs.,
* with neurogenic orthostatic hypotension associated with primary autonomic failure (Parkinson Disease, Multiple System Atrophy and Pure Autonomic Failure). Orthostatic hypotension will be defined as ≥20 mmHg decrease in systolic BP or ≥10 mmHg of diastolic BP within 3 minutes on standing associated with impaired autonomic reflexes determined by autonomic testing in the absence of other identifiable causes (Freeman et al., 2011).
* Patients able and willing to provide informed consent.

Exclusion Criteria:

* Pregnancy.
* Significant cardiac, renal or hepatic illness, or with contraindications to administration of pressor agents or external abdominal compression will be excluded.
* Clinically unstable coronary artery disease, or major cardiovascular or neurological event in the past 6 months, and; other factors which in the investigator's opinion would prevent the subject from completing the protocol including clinically significant abnormalities in clinical, mental or laboratory testing

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2015-04 (Actual); Primary Completion 2026-11-15 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Stroke volume | an average of 15 minutes of head up tilt
  Percent change from supine in stroke volume during head up tilt

SECONDARY OUTCOMES:
Systolic blood pressure | an average of 15 minutes of head up tilt
  Change from baseline in systolic blood pressure during head up tilt
Splanchnic vascular volume | an average of 15 minutes of head up tilt
  Percent change from supine in splanchnic vascular volume during head up tilt.

CONTACTS AND LOCATIONS:
Overall Officials: Italo Biaggioni, MD, Principal Investigator — Vanderbilt University; Luis E Okamoto, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No